CLINICAL TRIAL: NCT03853551
Title: A Prospective, Multicenter, Phase-IV Clinical Trial to Assess Safety of Osimertinib in Indian Adult Patients With Metastatic Epidermal Growth Factor Receptor (EGFR) T790M Mutation-positive Non-small Cell Lung Cancer (NSCLC).
Brief Title: Osimertinib Study in Indian Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5161C00005
Record Dates: First submitted 2019-02-20; First posted 2019-02-25 (Actual); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
Keywords: Non small cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single (Experimental): Single arm
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Osimertinib is an oral, potent, selective, irreversible inhibitor of both epidermal growth factor receptor - Tyrosine kinase inhibitors (EGFR-TKI) sensitizing and resistance mutations in nonsmall cell lung cancer (NSCLC) with a significant selectivity margin over wild-type EGFR.

SUMMARY:
This is a prospective, single-arm, multicenter, phase-IV study investigating the safety of osimertinib in Indian adult patients.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multicenter, phase-IV trial investigating the safety of osimertinib in Indian adult patients with locally advanced or metastatic EGFR-T790M mutation-positive NSCLC.

Prior to data collection, all patients must sign an informed consent form (ICF) allowing data collection and source data verification in accordance with local requirements and sponsor policy.

Patients with metastatic EGFR T790M mutation-positive NSCLC, who are eligible to osimertinib treatment as per locally approved prescribing information and ratified by an independent clinical judgment of treating physician will be evaluated for the inclusion into the current phase-IV study based on eligibility criteria. EGFR T790M positivity on plasma or tissue biopsy on PCR-based platform will be considered appropriate test. EGFR T790M must be performed after progressive disease on last line of therapy (on or after EGFR TKI therapy). In order to enroll approximately 60 patients, it is expected that approximately 70 patients will be screened.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of either gender and ≥18 years of age
2. Patients with metastatic EGFR T790M mutation-positive NSCLC, as detected by an appropriate test, who have progressed on or after EGFR TKI therapy by an independent clinical judgment of treating physician based on locally approved prescribing information
3. Each patient must sign an informed consent form (ICF)

Exclusion Criteria:

1. Patient with either the history of hypersensitivity to excipients of the study drug or to drugs with a similar chemical structure or class to the study drug.
2. Pregnant and/or lactating women
3. Patients participating in any current or future interventional trial will not be enrolled in the current study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- India (5):
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, New Dehli
  - Research Site, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Malik PS, Noronha V, Dabkara D, Maddu VK, Rajappa S, Limaye S, Batra U. Safety of osimertinib in adult patients with metastatic epidermal growth factor receptor T790M mutation-positive non-small cell lung cancer: Results from a Phase IV study in India. Indian J Cancer. 2022 Mar;59(Supplement):S1-S10. doi: 10.4103/ijc.ijc_1374_21. PMID 35343187
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5161C00005&attachmentIdentifier=e93b260a-ef33-4962-a0dc-98e6920b0420&fileName=D5161C00005_Redacted_CSP.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5161C00005&attachmentIdentifier=2db171c2-5c3c-47ff-b6ad-243f940f9ff4&fileName=D5161C00005-Redacted_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, open label, single arm, multicentre, India-specific Phase 4 study to investigate the safety of osimertinib 80 mg tablet in Indian adults with metastatic epidermal growth factor receptor (EGFR) T790M mutation positive non small cell lung cancer (NSCLC).
  60 Indian subjects were enrolled into the study.
Groups:
- Single Arm: single arm, open label study and Osimertinib 80 mg tablet was given orally once daily.
Period: Overall Study
Arm/Group | Single Arm
Started (60 patients were enrolled and received at least 1 dose of the study drug.) | 60
Completed (51 patients completed the study treatment (Cycle 1, Day 1 to Cycle 6, Day 21) and 28 days follow-up. Each cycle consisting of 21 days.) | 51
Not Completed | 9
Not completed — Death | 2
Not completed — 7 patients discontinued the study because of disease progression. | 7

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: Years] | 58 [34 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Only Indian) | 60

OUTCOME MEASURES:

1. Primary Outcome: Safety of Osimertinib
Description: Number of Patients with treatment emergent Adverse Events
Time Frame: 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 60
Participants | 60

ADVERSE EVENTS:
Time Frame: 6 months
Description: An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 3/60
Serious Adverse Events (participants affected / at risk) | 7/60
Other Adverse Events (participants affected / at risk) | 51/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=60)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cataract (Eye disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Mouth Ulceration (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1)
Disease progression (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=60)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 6 (7)
Decreased appetite (General disorders) | 5 (5)
Mucosal inflammation (General disorders) | 4 (4)
Paronychia (Infections and infestations) | 4 (5)
Blood creatine phosphokinase increased (Investigations) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution and/or investigator/Physician or Sponsor will provide a copy of any proposed publication or presentation for review and comment at least sixty (60) days prior to submission for publication.

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT03853551/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT03853551/SAP_001.pdf